CLINICAL TRIAL: NCT06248346
Title: Association Between Administration of Dexmedetomidine and Postoperative Mortality in Hospitals Among Inpatients Undergoing Surgeries Under General Anaesthesia Using Propofol
Brief Title: Association Between Administration of Dexmedetomidine and Postoperative Mortality in Hospitals
Status: Completed | Type: Observational
Sponsor: Xijing Hospital (Other)
Collaborators: The Affiliated Hospital of Qingdao University (Other); First Hospital of China Medical University (Other); The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School (Other); Sir Run Run Shaw Hospital (Other)
Responsible Party: Principal Investigator, Chong Lei, MD & phD, Principal Investigator, Xijing Hospital
Other Study IDs: KY20192045-C-1
Record Dates: First submitted 2024-01-24; First posted 2024-02-08 (Actual); Last update posted 2024-02-08 (Actual); Status verified 2024-01

CONDITIONS: In-hospital Mortality
MeSH Terms: interventions — Dexmedetomidine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- dexmedetomidine: dexmedetomidine group: abbreviated for dexmedetomidine group, refers to the group with intraoperative administration of dexmedetomidine adjunct to propofol
  Interventions: Drug: Dexmedetomidine
- non-dexmedetomidine: non-dexmedetomidine group: abbreviated for non-dexmedetomidine group, refers to the group without intraoperative administration of dexmedetomidine adjunct to propofol

INTERVENTIONS:
Drug: Dexmedetomidine — whether intraoperative dexmedetomidine was administered adjunct to propofol for patients undergoing surgeries under general anaesthesia
  Groups: dexmedetomidine

SUMMARY:
The present multicentre retrospective cohort study aimed to investigate the association between intraoperative administration of dexmedetomidine and postoperative mortality in hospitals.

The investigators set out to test the hypothesis that perioperative dexmedetomidine use, as an adjunct to general anesthesia, diminishes postoperative mortality in hospitals across all categories of surgical patients.

ELIGIBILITY:
Inclusion Criteria:

* adult patients (aged ≥18 years)
* undergo general anaesthesia with propofol
* from January 1, 2014 to June 30, 2018

Exclusion Criteria:

* patients undergoing intervention procedures under monitored anaesthesia care (MAC)
* patients undergoing minor procedures under local or regional anaesthesia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All adult patients (aged ≥18 years) admitted for surgical procedures under general anaesthesia with propofol at the five participating hospitals from January 1, 2014 to June 30, 2018.
Sampling Method: Non-Probability Sample
Enrollment: 518043 (Actual)
Dates: Start 2014-09-01 (Actual); Primary Completion 2018-06-30 (Actual); Study Completion 2018-07-01 (Actual)

PRIMARY OUTCOMES:
in-hospital all-cause mortality | from the time of end of surgery until time of documented hospital discharge or time of death, whichever came first, assessed up to 1 year
  in-hospital deaths or discharged to hospice (or home)

SECONDARY OUTCOMES:
length of postoperative hospital stay | from the time of end of surgery until time of documented hospital discharge or time of death, whichever came first, assessed up to 1 year
  in days
admission to the intensive care unit (ICU) | from the time of end of surgery until time of documented hospital discharge or time of death, whichever came first, assessed up to 1 year
  unplanned admissions
adverse events after surgery | from the time of end of surgery until time of documented hospital discharge or time of death, whichever came first, assessed up to 1 year
  severe stroke, the necessity for renal replacement therapy (RRT), myocardial infarction, ventilator-associated pneumonia (VAP), acute respiratory distress syndrome (ARDS), unplanned reoperation due to postoperative complications, sepsis, and multi-organ dysfunctions (MODs), if any

IPD SHARING:
Plan to Share IPD: No
IPD will not be available